CLINICAL TRIAL: NCT07140783
Title: RANDOMIZED, PLACEBO-CONTROLLED, DOUBLE-MASKED STUDY OF THE SAFETY AND EFFICACY OF POS (0.75% PHENTOLAMINE OPHTHALMIC SOLUTION) IN PARTICIPANTS WITH PREVIOUS KERATOREFRACTIVE SURGERY WITH DECREASED VISUAL ACUITY UNDER MESOPIC CONDITIONS
Brief Title: OPI-NXYDLD-303 Safety and Efficacy of Phentolamine Ophthalmic Solution in Keratorefractive Surgery Participants With Decreased Mesopic Visual Acuity
Acronym: LYNX-3
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ocuphire Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OPI-NYXDLD-303 (LYNX-3)
Record Dates: First submitted 2025-08-22; First posted 2025-08-26 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Vision Loss Night; Vision Disorders
Keywords: keratorefractive surgery; decreased visual acuity; vision disorder; mesopic lighting; night vision
MeSH Terms: conditions — Vitamin A Deficiency; Vision Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 0.75% Phentolamine Ophthalmic Solution (Experimental): 0.75% Phentolamine Ophthalmic Solution
  Interventions: Drug: 0.75% Phentolamine Ophthalmic Solution
- Placebo - Phentolamine Ophthalmic Solution vehicle (Placebo Comparator): Placebo-phentolamine ophthalmic solution vehicle
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 0.75% Phentolamine Ophthalmic Solution — Once daily dosing
  Other Names: phentolamine ophthalmic solution 0.75%, a non-selective alpha-1 and alpha-2 adrenergic antagonist
  Arms: 0.75% Phentolamine Ophthalmic Solution
Drug: Placebo — Once daily dosing
  Other Names: POS vehicle placebo
  Arms: Placebo - Phentolamine Ophthalmic Solution vehicle

SUMMARY:
The goal of this clinical trial is to learn if Phentolamine Ophthalmic Solution works to treat adults that have had keratorefractive surgery and have decreased visual acuity under mesopic conditions. It will also learn about the safety of Phentolamine Ophthalmic Solution. The main questions it aims to answer are:

Researchers will compare Phentolamine Ophthalmic Solution to a placebo (a look-alike substance that contains no drug) to see if Phentolamine Ophthalmic Solution works to improve vision in low light conditions.

Participants will:

Take Phentolamine Ophthalmic Solution or a placebo drop every day for 2 weeks Visit the clinic once every week for 2 weeks for checkups and tests Keep a diary of when they instill the study medication each evening

DETAILED DESCRIPTION:
OPI-NXYDLD-303 RANDOMIZED, PLACEBO-CONTROLLED, DOUBLE-MASKED STUDY OF THE SAFETY AND EFFICACY OF POS (0.75% PHENTOLAMINE OPHTHALMIC SOLUTION) IN PARTICIPANTS WHO HAVE PREVIOUSLY HAD KERATOREFRACTIVE SURGERY AND HAVE DECREASED VISUAL ACUITY UNDER MESOPIC CONDITIONS

ELIGIBILITY:
Inclusion Criteria:

1. Males or females ≥ 18 years of age
2. Previous history (>6 months prior to Screening) of keratorefractive surgery (eg, PRK, LASIK, SMILE, and RK/astigmatic keratotomy [AK]/limbal-relaxing incisions [LRI]) in one or both eyes and have participant-reported night vision disturbances (eg, glare, halos, and/or starbursts). Symptoms must have been first noted within 2 months following keratorefractive surgery
3. Able to independently comply with all protocol-mandated procedures and to attend all scheduled office visits
4. Able and willing to give written consent to participate in this study
5. Able to self-administer study medication

   Inclusion criteria #6, #7, and #8 must all be met in the same eye:
6. PD ≥ 5 mm under mesopic conditions in at least 1 eye. This test may be repeated once, following an additional 5 min of dark adaptation to the mesopic light conditions if the initial results do not meet this criterion
7. mLCVA ≤ 30 Early Treatment Diabetic Retinopathy Study (ETDRS) letters (20/63 Snellen or worse) in at least 1 eye using the Precision Vision Illuminator Cabinet with 5% translucent contrast chart and a mesopic filter at 4 m
8. ≥ 10 ETDRS letters improvement in mLCVA in at least 1 eye during illumination of the contralateral eye with a Brightness Acuity Tester (BAT) system on the low setting using the Precision Vision Illuminator Cabinet with 5% translucent contrast chart and a mesopic filter at 4 m

Exclusion Criteria:

Ophthalmic (in either eye unless otherwise noted):

1. Prior unresolved dry eye diagnosis, taking prescription medication for dry eye (eg, drops, nasal sprays [Tyrvaya®], etc.), or taking artificial tear drops routinely for dry eye
2. Prior history of fluctuating vision
3. Clinically significant ocular disease as deemed by the Investigator (eg, untreated visually significant cataract, glaucoma, corneal edema, uveitis, severe keratoconjunctivitis sicca, retina degeneration, loss of visual field due to glaucoma or stroke, branch retinal vein occlusion, retina flare) that might interfere with the study
4. History or presence of corneal endothelial dystrophy (eg, Fuchs' dystrophy or presence of guttae)
5. Known hypersensitivity to any topical alpha-adrenoceptor antagonists
6. Known allergy or contraindication to any component of the vehicle formulation
7. History of cauterization of the punctum or punctal plug (silicone or collagen) insertion or removal in the study eye
8. Pseudophakic participants with extended depth-of-focus or multifocal intraocular lenses (IOLs)
9. Ocular trauma, ocular surgery (eg, IOLs), or laser procedure (eg, LASIK, PRK, SMILE, and RK/AK/LRI) within 6 months prior to Screening
10. Use of any topical prescription or over-the-counter (OTC) ophthalmic medications of any kind (including artificial tear drops) within 7 days prior to Screening until study completion, with the exception of lid scrubs with OTC products (eg, OCuSOFT® lid scrub, SteriLid®, baby shampoo, etc.)
11. Recent or current evidence of ocular infection or inflammation (such as current evidence of clinically significant blepharitis, conjunctivitis, or a history of herpes simplex keratitis or herpes zoster keratitis at Screening). Participants must be symptom free for at least 7 days prior to Screening
12. History of diabetic retinopathy, diabetic macular edema, or dry or wet macular degeneration in the study eye
13. History of any traumatic (surgical or nonsurgical) or nontraumatic condition affecting the pupil or iris (eg, irregularly shaped pupil, neurogenic pupil disorder, iris atrophy, iridotomy, iridectomy, etc.)
14. Unwilling or unable to discontinue use of contact lenses at least 1 hour prior to Screening for soft contact lenses or at least 8 hours prior to Screening for hard gas-permeable contact lenses, and at least 8 hours (for both types of lenses) prior to all other office visits
15. Previously undiagnosed dry eye, at the determination of the Investigator. Dry eye diagnosis should be based on one of the following dry eye test results: tear break-up time < 5 seconds, or corneal fluorescein staining ≥ Grade 2 in the inferior zone or ≥ Grade 1 in the central zone using the National Eye Institute scale

    Systemic:
16. Known hypersensitivity or contraindication to alpha- and/or beta-adrenoceptor antagonists
17. Clinically significant systemic disease (eg, severe diabetes, myasthenia gravis, cancer, hepatic, renal, endocrine, or cardiovascular disorders) that might interfere with the study
18. Initiation of treatment with or any changes to the current dosage, drug, or regimen of any systemic adrenergic or cholinergic drugs within 7 days prior to Screening or during the study
19. Participation in any investigational study within 30 days prior to Screening or during the study
20. Participation in any investigational study using POS
21. Females of childbearing potential who are pregnant, nursing, planning a pregnancy during the study, or not using a medically acceptable form of birth control. Acceptable methods include the use of at least one of the following: intrauterine device, hormonal contraception (oral, injection, patch, implant, ring), barrier with spermicide (condom, diaphragm), or abstinence. A female is considered to be of childbearing potential unless she is 1 year postmenopausal or 3 months post-surgical sterilization. All females of childbearing potential, including those post-tubal ligation, must have a negative urine pregnancy test result at each visit
22. Resting HR outside 50 to 110 beats per min at Screening. HR may be repeated only once if outside the specified range, following at least a 5-min rest period in the sitting position
23. Hypertension with resting diastolic BP > 105 mmHg or systolic BP > 160 mmHg at Screening. BP may be repeated only once if outside the specified range, following at least a 5-min rest period in the sitting position

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-09-02 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Percent of participants with >= 15 ETDRS letters (>= 3 lines) improvement in the study eye in mLCVA compared to Baseline (Day1 pre-dose) at Day 15 | Day 15
  To evaluate the efficacy of POS to improve mLCVA in subjects with previous keratorefractive surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jay Pepose, MD, Study Chair — Opus Genetics/Ocuphire Pharma
Locations (23):
- United States (23):
  - Arizona Eye Care, Chandler, Arizona
  - Carrot Eye Center, Mesa, Arizona
  - Eye Doctors of Arizona, Phoenix, Arizona
  - MRB Eye Care Consultants, Scottsdale, Arizona
  - Global Research Management, Glendale, California
  - Gordon Schanzlin New Vision, La Jolla, California
  - Eye Research Foundation, Newport Beach, California
  - California Eye Specialists Medical Group, Pasadena, California
  - NVISION Clinical Research, San Diego, California
  - Scripps Poway Eyecare and Optometry, San Diego, California
  - Wolsten and Goldberg Eye Assoc., Torrance, California
  - Glaucoma Specialist of South Florida, Delray Beach, Florida
  - Segal Drug Trials, Delray Beach, Florida
  - Wyse Eyecare, Northbrook, Illinois
  - Virdi Eye Clinic, Rock Island, Illinois
  - Durrie Vision, Overland Park, Kansas
  - Kannarr Eye Care, Pittsburg, Kansas
  - Eye Health Vision Center, South Dartmouth, Massachusetts
  - Northeast Eye Research Associates, Woburn, Massachusetts
  - Oculus Research, Garner, North Carolina
  - West Bay Eye Assoc., Warwick, Rhode Island
  - Zillan Clinical Research, Houston, Texas
  - Hoopes Vision, Draper, Utah

IPD SHARING:
Plan to Share IPD: No